CLINICAL TRIAL: NCT05737017
Title: A Randomized Active-controlled Clinical Trial to Investigate the Efficacy and Safety of a Hybrid Hemostatic Device (ClearCoajet) During Endoscopic Resection for Colorectal Tumors
Brief Title: The Efficacy and Safety of a Hybrid Hemostatic Device (ClearCoajet)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Han Hee Lee, Associate Professor, Yeouido St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Coajet_LGI
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The ClearCoajet group (Experimental): During the endoscopic resection procedures, the ClearCoajet will be used for injection and initial hemostasis for intraprocedural bleeding.
  Interventions: Device: ClearCoajet
- The control group (Active Comparator): During the endoscopic resection procedures, the conventional injector will be used for injection.
  Interventions: Device: ClearCoajet

INTERVENTIONS:
Device: ClearCoajet — The ClearCoajet is a new hemostasis device with a hybrid function (Coagulation + Injection) and is developed to provide effective coagulation, injection, and marking around lesions without changing devices during the endoscopic procedure.

SUMMARY:
The ClearCoajet is a new hemostasis device with a hybrid function (Coagulation + Injection) and is developed to provide effective coagulation, injection, and marking around lesions without changing devices during the endoscopic procedure. In this study, the investigators examine the hemostatic effect of ClearCoajet on intraprocedural bleeding during endoscopic mucosal resection or endoscopic submucosal dissection for colorectal sessile polyps or lateral growth tumors larger than 1.5 cm. The investigators also aim to compare the delayed bleeding and recurrence rates between the ClearCoajet group and the control group.

ELIGIBILITY:
Inclusion Criteria:

* patients with colorectal sessile polyps or lateral growth tumors larger than 1.5 cm

Exclusion Criteria:

* Pedunculated polyp
* Patients with coagulopathy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemostasis of intraprocedural bleeding | during endoscopic resection for colorectal lesions
  Hemostasis efficacy of intraprocedural bleeding during endoscopic resection for colorectal lesions

SECONDARY OUTCOMES:
Delayed bleeding rate | within 4 weeks after endoscopic resection
  Delayed bleeding rate within 4 weeks after endoscopic resection
Complication rate | within 4 weeks after endoscopic resection
  Complication rate

CONTACTS AND LOCATIONS:
Locations (1):
- Yeouido St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided